CLINICAL TRIAL: NCT03415308
Title: Development and Pilot Testing of an Implicit Bias Training Intervention for Providers to Advance Equity in Healthcare
Brief Title: REACH Implicit Bias Training Project
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00088354
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Communication; Bias, Racial; Relation, Doctor Patient
Keywords: Implicit Bias; Healthcare Equity
MeSH Terms: conditions — Communication; Racism; Bias, Implicit | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient Focus Groups: Identify patient preferences for constructs, and related outcomes, that reflect the expression of implicit bias in clinical encounters. I
  Interventions: Other: Focus Groups
- Stakeholders Cognitive Interviews: Investigators will conduct a series of semi-structured interviews.
  Interventions: Other: Cognitive Interviews
- Pilot Testing of Implicit Bias Training: Refined intervention emerging from Aim 2. T
  Interventions: Other: Pilot Testing of Implicit Bias Training

INTERVENTIONS:
Other: Focus Groups — Investigators will use qualitative methods to gather data on the elements associated with the patient perception of implicit bias (e.g. communication, respect, patient-centeredness) to ensure that our selected outcomes reflect the breadth of patients' concerns.
  Groups: Patient Focus Groups
Other: Cognitive Interviews — To gather insights from stakeholders regarding how to best refine the design of our existing implicit bias intervention to ensure that we have addressed potential facilitators and barriers to uptake, use, and sustainability
  Groups: Stakeholders Cognitive Interviews
Other: Pilot Testing of Implicit Bias Training — Determine the feasibility of delivering the refined implicit bias reduction intervention and assessing patient centered outcomes by giving providers a refined implicit bias training.
  Groups: Pilot Testing of Implicit Bias Training

SUMMARY:
The overall goal and theme of the Duke Center for Research to Advance Equity in Healthcare is to reduce racial and ethnic disparities in health through interventions that affect the clinical encounter. To achieve this goal, there is an urgent need for interventions that address implicit bias in healthcare. Implicit bias training is widely used to raise self-awareness and provide self-management tools. The overall objective is to test the hypothesis that implicit bias training for healthcare providers will reduce racial and ethnic disparities in patient- centered care. The proposed project will lay the groundwork for testing that hypothesis by using patient focus groups to garner a deeper understanding of perceptions of implicit bias in the clinical encounter; provider and health system stakeholder semi-structured interviews to inform refinement of the existing implicit bias training at Duke; and perform a pilot study of implicit bias training for providers. At the conclusion of this study, the investigators will have the necessary preliminary data to propose a definitive trial to determine the impact of an implicit bias training intervention for providers on racial and ethnic disparities in patient-centered care. This research will ultimately lead to the delivery of equitable, evidence-based, patient-centered care for all.

DETAILED DESCRIPTION:
Despite substantial improvements in the overall health of our nation, racial and ethnic disparities in health and healthcare remain ubiquitous. Disparities are apparent after controlling for access to care, insurance, income, patient preferences, and clinical need, suggesting that providers and health systems are important contributors to racial disparities in healthcare. In its landmark report, "Unequal Treatment," the Institute of Medicine concluded that providers contribute to disparities through the effects of implicit bias. Implicit bias occurs when thoughts and feelings outside of conscious awareness and control affect judgment and/or behavior. It is closely related to stereotyping, but not necessarily associated with explicit bias (i.e., prejudice). It leads to involuntary "blind spots" in virtually all of us. Implicit racial bias in providers is associated with Blacks (compared to Whites) experiencing lower patient-centered communication, worse doctor-patient relationships, lower confidence in the doctor, and poorer health outcomes. Therefore, to address health disparities, there is an urgent need for interventions that address implicit bias in healthcare.

Across society, implicit bias training is increasingly used in public service, business and healthcare settings to raise self-awareness and provide self-management tools for avoiding actions based on implicit bias. While such interventions are well-conceived and intuitively attractive, they have not been rigorously tested. In order to make optimal use and insure sustained support for such training, its effectiveness must be rigorously demonstrated. The overall objective is to test the hypothesis that implicit bias training for healthcare providers will reduce racial/ethnic disparities in patient-centered care. Before investigators can definitively test this hypothesis, additional groundwork must be done.

This project will provide the preliminary evidence necessary to ultimately evaluate an implicit bias training intervention in a pragmatic, randomized clinical trial conducted at the health system level. To do so, investigators will achieve these specific aims:

Aim 1. Identify patient preferences for constructs, and related outcomes, that reflect the expression of implicit bias in clinical encounters. Investigators will use qualitative methods to gather data on the elements associated with the patient perception of implicit bias (e.g. communication, respect, patient-centeredness) to ensure that our selected outcomes reflect the breadth of patients' concerns.

Aim 2. Refine an existing implicit bias intervention with input from providers, health system stakeholders and expert consultation. Investigators will conduct a series of semi-structured interviews to gather insights from stakeholders regarding how to best refine the design of our existing implicit bias intervention to ensure that we have addressed potential facilitators and barriers to uptake, use, and sustainability.

Aim 3. In a pilot trial, determine the feasibility of delivering the refined implicit bias reduction intervention and assessing patient centered outcomes. Investigators will conduct a feasibility trial using the refined intervention emerging from Aim 2. These feasibility outcomes will prepare investigators for a future, fully-powered randomized trial of implicit bias training.

At the conclusion of this study, investigators will be prepared to test the impact of implicit bias training on racial/ethnic disparities in the clinical encounter, and thus move us toward delivery of equitable, evidence-based, patient- centered clinical care.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

* Had at least 2 non-urgent ambulatory care visits any Healthcare facility in the past year (via self-report)
* Proficient in English

Aim 2:

* Providers from Durham-based ambulatory clinics in the Duke Health System or Stakeholder

Aim 3:

* Providers from the Duke Health System providing care to a continuity patient panel.

Exclusion Criteria:

Aim 1:

* Less than 2 non-urgent visits
* Patient not identifying as black, white or Hispanic
* Non-English speaking

Aim 2:

* Not a Duke provider or stakeholder

Aim 3:

* Not a Duke Health system provider/affiliated provider
* Does not provide clinical care at a Duke affiliated facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For Aim 1, investigators will use the community population. Aims 2 and 3 focus specifically on providers and stakeholders at Duke medical center.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary G Bennett, Ph.D, Principal Investigator — Duke University; Kimberly S Johnson, MD, Study Director — Duke University; Laura P Svetkey, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Svetkey LP, Bennett GG, Reese B, Corsino L, Pinheiro SO, Fischer JE, Seidenstein J, Olsen MK, Brown T, Ezem N, Liu E, Majors A, Steinhauser KE, Sullivan BH, van Ryn M, Wilson SM, Yang H, Johnson KS. Design and pilot test of an implicit bias mitigation curriculum for clinicians. Front Med (Lausanne). 2024 Jun 6;11:1316475. doi: 10.3389/fmed.2024.1316475. eCollection 2024. PMID 38903809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Focus Groups | Stakeholders Cognitive Interviews | Pilot Testing of Implicit Bias Training
Started | 50 | 27 | 37
Completed | 50 | 27 | 29
Not Completed | 0 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Scheduling Conflicts | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Focus Groups | Stakeholders Cognitive Interviews | Pilot Testing of Implicit Bias Training | Total
Number analyzed (Participants) | 50 | 27 | 37 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected from providers in Aim 2 and Aim 3.
  years
    number analyzed (Participants) | 50 | 0 | 0 | 50
    (all) | 42.4 (15.9) |  |  | 42.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 16 | 29 | 85
  Male | 10 | 11 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 1 | 1 | 13
  Not Hispanic or Latino | 39 | 11 | 36 | 86
  Unknown or Not Reported | 0 | 15 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 10 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 20 | 8 | 2 | 30
  White | 26 | 18 | 24 | 68
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 4 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Training Measured by Participation
Description: Investigators will judge the trial as feasible if at least 50% of eligible providers agree to participate.
Time Frame: 4 hours (post-training)
Population: Data not collected.
Arm/Group | Patient Focus Groups | Stakeholders Cognitive Interviews | Pilot Testing of Implicit Bias Training
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Acceptability
Description: At least 80% of those enrolled complete the trial (attend both sessions); and achieve at least 75% adherence to all intervention activities and exercises.
Time Frame: 4 hours (post-training)
Population: Primary outcome was only measured for participants enrolled in Aim 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Focus Groups | Stakeholders Cognitive Interviews | Pilot Testing of Implicit Bias Training
Number analyzed (Participants) | 0 | 0 | 37
Participants |  |  | 29

3. Secondary Outcome: Variability in Any Trial Outcomes by Provider-related Characteristics
Description: Investigators will also gather provider data (age, sex, race, practice characteristics, time in practice, etc.) via self-report and assess and variability in outcomes by these characteristics.
Time Frame: 4 hours (post-training)
Population: Data not collected.
Arm/Group | Patient Focus Groups | Stakeholders Cognitive Interviews | Pilot Testing of Implicit Bias Training
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in IAT Outcomes From Baseline to Immediately Post-intervention
Description: Investigators will ask participants to complete an implicit association test (IAT) at baseline and immediately following training using the Brief IAT measure, which can be administered in under 5 minutes on a laptop computer. The Brief IAT provides comparable findings on implicit racial attitudes tests, when validated against the longer IAT measure.
Time Frame: baseline, 4 hours (post-training)
Population: Data not collected.
Arm/Group | Patient Focus Groups | Stakeholders Cognitive Interviews | Pilot Testing of Implicit Bias Training
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 hours (post-training)
Arm/Group | Patient Focus Groups | Stakeholders Cognitive Interviews | Pilot Testing of Implicit Bias Training
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/27 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/27 | 0/37
Other Adverse Events (participants affected / at risk) | 0/50 | 0/27 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03415308/Prot_ICF_000.pdf